CLINICAL TRIAL: NCT01337271
Title: Performance of Neurally Adjusted Ventilatory Assist (NAVA) During an Spontaneous Breathing Trial
Brief Title: Performance of Neurally Adjusted Ventilatory Assist (NAVA) During Spontaneous Breathing Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: 2010-345
Record Dates: First submitted 2011-04-12; First posted 2011-04-18 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Respiratory Failure
Keywords: artificial, ventilation; mechanical ventilation; weaning
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- PSV (Active Comparator)
  Interventions: Procedure: SBT- PSV; Procedure: SBT - NAVA
- NAVA (Experimental)
  Interventions: Procedure: SBT- PSV; Procedure: SBT - NAVA

INTERVENTIONS:
Procedure: SBT- PSV — An Spontaneous breathing trial for 30 minutes on pressure support ventilation, which is a commonly used strategy to evaluate readiness for extubation
  Other Names: SBT
Procedure: SBT - NAVA — An spontaneous breathing trial (SBT) on the ventilatory mode NAVA, with ventilatory support titrated to be similar to the support provided during an SBT on pressure support mode (PSV). NAVA captures the electrical activity of the diaphragm with an esophageal-gastric catheter, and uses the electrical signal to deliver inspiratory pressure proportional to the intensity of patient effort, as well as to trigger and cycle assisted mechanical breaths.
  Other Names: NAVA; N.A.V.A.

SUMMARY:
The purpose of this study is to compare a new mode of mechanical ventilation (NAVA, or Neurally adjusted Ventilatory assist) with a traditional mode (Pressure Support ventilation) on its the ability to detect patients ready for extubation (liberation from mechanical ventilation).

DETAILED DESCRIPTION:
Patients under mechanical ventilation who are suspected to be recovered and ready to return to spontaneous ventilation often undergo an spontaneous breathing trial (SBT) before extubation and liberation from mechanical ventilation. During the test, which lasts from 30 minutes to 2 hours , the patient receives minimal support from the ventilator, and the ICU team observes if the patient develops any signs or symptoms of discomfort or respiratory distress. If the patient tolerates the test, he or she is considered ready for extubation. The Neurally Adjusted Ventilatory Assist (NAVA) is a new mode of ventilation, shown to improve patient-ventilator synchrony. It has not been tested during SBTs. Our objective is to compare the performance of NAVA with the commonly used Pressure Support ventilation, during an SBT. Patients considered to be ready for an SBT by the ICU team will undergo two SBTs in random order: one in pressure support, and the other on NAVA, with a 1-hour interval between the tests. Ventilatory parameters and patient-ventilator interaction variables will be compared among the two tests.

This study will help us understand if NAVA can be used during an SBT, which might be important for patients who are being ventilated with NAVA before the SBT is suggested, especially those how present a high asynchrony rate when ventilated with Pressure Support Mode.

ELIGIBILITY:
Inclusion Criteria:

* mechanical ventilation for more than 48 hours
* Considered ready for an spontaneous breathing trial by the ICU team
* informed consent for participation on the study signed by a family member

Exclusion Criteria:

* age < 18yrs
* pregnancy
* facial trauma or burns that might interfere with the esophageal catheter placement
* nasal pathologies that prevent adequate placement of the catheter
* esophageal varices or gastroesophageal bleeding in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
rate of success on the spontaneous breathing trial | 30 minutes, or earlier (if the SBT is interrupted for intolerance), i.e., at the end of the spontaneous breathing trial
  The ICU team will observe the patient during the spontaneous breathing trial, and use standard objective (blood gases) and subjective (including respiratory rate, tidal volume, comfort, hemodynamic variables) variables to determine if the patient tolerates the SBT and therefore is ready for discontinuation from mechanical ventilation

SECONDARY OUTCOMES:
Extubation failure rate | 48 hours after extubation
  Patients who are extubated within 24 hours of the completion of the study will be followed for 48h, and if re-intubation is required within these first 48h after the extubation, the investigators will consider that the patient had extubation failure

CONTACTS AND LOCATIONS:
Overall Officials: Juliana C Ferreira, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Respiratory ICU, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Ferreira JC, Diniz-Silva F, Moriya HT, Alencar AM, Amato MBP, Carvalho CRR. Neurally Adjusted Ventilatory Assist (NAVA) or Pressure Support Ventilation (PSV) during spontaneous breathing trials in critically ill patients: a crossover trial. BMC Pulm Med. 2017 Nov 7;17(1):139. doi: 10.1186/s12890-017-0484-5. PMID 29115949